CLINICAL TRIAL: NCT07271264
Title: A Randomised Paired Design Study of Texture and Colour Enhancement Imaging (TXI) Versus High-definition White Light Endoscopy for Dysplasia Detection in IBD Surveillance.
Brief Title: A Randomised Paired Design Study of Texture and Colour Enhancement Imaging (TXI) Versus High-definition White Light Endoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD25/051
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: IBD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TXI (Active Comparator): Participants allocated to the "TXI" group undergo withdrawal using Texture and Colour Enhancement Imaging
  Interventions: Diagnostic Test: TXI
- White light (Other): Participants allocated in the "White light " group receive withdrawal with White light
  Interventions: Diagnostic Test: TXI

INTERVENTIONS:
Diagnostic Test: TXI — Participants allocated to the "TXI" group undergo withdrawal using Texture and Colour Enhancement Imaging, while those in the "white light" group receive withdrawal with with high-definition white light endoscopy. Both procedures follow standardized protocols outlined in the study design.

SUMMARY:
Texture and Colour Enhancement Imaging (TXI) improves texture, brightness, and colour in white-light endoscopy to highlight subtle tissue differences. Now available through the EVIS X1 system, early evidence suggests potential value in IBD. Studies show that TXI may help predict ulcerative colitis relapse and performs comparably to dye chromoendoscopy in detecting lesions, though no randomised data exist for dysplasia detection in IBD surveillance. We therefore propose a randomised paired study comparing TXI with high-definition white-light endoscopy for dysplasia detection in IBD surveillance.

DETAILED DESCRIPTION:
Texture and colour enhancement imaging (TXI) is designed to enhance texture, brightness and colour in white light in order to clearly define subtle tissue differences. This has been shown to enhance subtle tissue differences (20). This technology has recently become available in routine clinical practice with introduction of the EVIS X1 system (Olympus). Some promising data about the use of TXI in IBD are emerging. In a prospective observational study, 146 UC patients in endoscopic remission were evaluated with WLE and TXI. Patients with accentuated redness and poor visibility of deep vessels at TXI had significantly lower UC relapse-free rates than patients with no redness or accentuated redness alone, suggesting a possible role of TXI in guiding treatment intensification (21). In a small study of 16 IBD patients undergoing surveillance colonoscopy, TXI missed no lesions detected by subsequent dye chromoendoscopy (22). There are no randomised data regarding the utility of TXI for detection of dysplasia in colonoscopy IBD surveillance. We propose to undertake a randomised paired design study of Texture and Colour Enhancement Imaging (TXI) versus high-definition white light endoscopy for dysplasia detection in IBD surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Patients >16 with inflammatory bowel disease undergoing surveillance colonoscopy.
* Patients with Crohn's (L2/L3 Montreal classification) with >50% colonic involvement OR
* Patients with ulcerative colitis with Extensive or left sided disease (E3 or E2 Montreal classification) for at least 8 years or a diagnosis of Primary sclerosing cholangitis concomitant with IBD.

Exclusion Criteria:

* Disease duration <8 years unless a diagnosis of PSC
* Incomplete colonoscopy
* BBPS <6 or <2 in any segment
* MES ≥2 or any variable of the SES-CD is ≥2 or any stenosis for >10cm segment (above the rectum)
* Previous colorectal resection
* Thrombocytopaenia (platelet count <50) or Coagulopathy precluding biopsy
* Anticoagulation that has not been held appropriately prior to the procedure (must be held at least the morning of the procedure).
* Pregnancy
* Unable or unwilling to consent to study participation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2028-12-08 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
To compare the proportion of patients with at least 1 dysplastic lesion detected using TXI compared with high-definition white light endoscopy. | 6 months
  The number of dysplastic areas detected during endoscopy

IPD SHARING:
Plan to Share IPD: No